CLINICAL TRIAL: NCT01031732
Title: A Prospective Randomized Controlled 4-arm Study for the Evaluation of 4 Surgical Techniques in Primary Total Hip Arthroplasty
Brief Title: Evaluation of Four Surgical Techniques in Primary Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Janet George/Director, Corporate External Research, Zimmer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-2177c
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Minimally invasive; Total hip arthroplasty; Functional outcome; To compare the surgical results of 4 MIS THA techniques; To investigate the functional outcomes of 4 MIS THA techniques; To study the biochemical parameters after the MIS surgeries.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Two-incision (Experimental): MIS-2 THA
  Interventions: Procedure: MIS-2 THA
- Watson-Jones (Experimental): MIS-WJ
  Interventions: Procedure: MIS-WJ
- MIS-AL (Experimental)
  Interventions: Procedure: MIS-AL THA
- MIS-PL (Experimental)
  Interventions: Procedure: MIS-PL THA

INTERVENTIONS:
Procedure: MIS-2 THA — MIS two-incision THA
  Arms: Two-incision
Procedure: MIS-WJ — MIS-Watson Jones THA
  Arms: Watson-Jones
Procedure: MIS-AL THA — Transgluteal approach
  Arms: MIS-AL
Procedure: MIS-PL THA — Posterolateral approach
  Arms: MIS-PL

SUMMARY:
Current "Minimally Invasive THR" includes: (1) Minimally Invasive Two-Incision THR (MIS-2), (2) Minimally Invasive Modified Watson-Jones THR (MIS-WJ). In contrast, "mini-incision" utilizes smaller incision (< 10 cm in definition) to perform the THR which can further be divided into mini-anterolateral (Mini-AL) and mini-posterolateral (Mini-PL).The purpose of this study is to investigate how MIS THR can affect the results of THR by a prospective randomized clinical trial. It is hoped that some new standards could be established for the total hip replacement surgery.

DETAILED DESCRIPTION:
The prospective randomized study will be performed in patients after obtaining patient's consent. "Envelop drawing based on random table" will decide the choice of approach. (1) Group 1: MIS-2, 30 cases (2) Group 2: MIS-WJ, 30 cases (3) Group 3: Mini-AL, 30 cases (4) Group 4: Mini-PL, 30 cases. Only the unilateral coxarthrosis will be recruited for the study. Analytical methods include (1) gait analysis (2) cybex study (3) balance test and obstacle crossing test (4) bone densitometry (5) PETS oxygen consumption and glucose utilization tests (6) inflammatory markers (7) clinical assessment (8) X-ray studies. Patients will be scheduled for specified examinations preoperatively, postoperatively and within 5 days, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip disease that is indicated for primary total hip arthroplasty.

Exclusion Criteria:

* A previous THA on the contralateral hip.
* Any condition contraindicated for primary total hip arthroplasty.
* Refuse to be randomized in the study arms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pain and Harris hip score | 5 days, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months

SECONDARY OUTCOMES:
Functional outcomes assessment | 6 weeks, 3 months, 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

REFERENCES:
- [Background] Chou SW, Ueng SW, Lee MS. Muscular recovery of hip flexors and extensors after two-incision total hip arthroplasty. Chang Gung Med J. 2008 Nov-Dec;31(6):576-82. PMID 19241897
- [Background] Chen DW, Hu CC, Chang YH, Yang WE, Lee MS. Comparison of clinical outcome in primary total hip arthroplasty by conventional anterolateral transgluteal or 2-incision approach. J Arthroplasty. 2009 Jun;24(4):528-32. doi: 10.1016/j.arth.2008.03.016. Epub 2008 Aug 3. PMID 18676112
- [Background] Hu CC, Yang WE, Chang YH, Chen DW, Ueng SW, Lee MS. Fluoroscopy cannot recognize intraoperative fracture in patients receiving 2-incision total hip arthroplasty. J Arthroplasty. 2008 Oct;23(7):1031-6. doi: 10.1016/j.arth.2007.09.026. Epub 2008 Mar 4. PMID 18534477
- [Background] Lu ML, Chou SW, Yang WE, Senan V, Hsieh PH, Shih HN, Lee MS. Hospital course and early clinical outcomes of two-incision total hip arthroplasty. Chang Gung Med J. 2007 Nov-Dec;30(6):513-20. PMID 18350734
- [Background] Lee MS, Kuo CH, Senan V, Chen WJ, Chen LH, Ueng SW. Two-incision total hip replacement: Intra-operative fluoroscopy versus imageless navigation for cup placement. Hip Int. 2006;16 Suppl 4:35-41. doi: 10.1177/112070000601604S08. PMID 19219827
- See also: Chang Gung Memorial Hospital — http://www.cgmh.org.tw
- See also: American Academy of Orthopaedic Surgeons — http://www.AAOS.org
- See also: Chang Gung University — http://www.cgu.edu.tw